CLINICAL TRIAL: NCT05215535
Title: Limerick - Liver Magnetic Resonance Imaging Before Treatment for Rectal Cancer. A Randomised Controlled Trial.
Brief Title: Liver Magnetic Resonance Imaging Before Treatment for Rectal Cancer. A Randomised Controlled Trial.
Acronym: Limerick
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Limerick
Record Dates: First submitted 2021-12-15; First posted 2022-01-31 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-05

CONDITIONS: Rectal Cancer
Keywords: rectal cancer; radiological examination liver
MeSH Terms: conditions — Rectal Neoplasms | interventions — Liver Extracts

STUDY DESIGN:
Intervention Model Description: Consenting patients with newly diagnosed rectal cancer who fulfil the inclusion criteria and no exclusion criteria will be randomized into two groups with regard to radiological investigation of the liver; Intervention: An abbreviated MRI of the liver/abdomen Control: A combined single venous and 3 min equilibrium phase CT of the abdomen/liver
  Randomization will be conducted in blocks of 6, and stratified for sex and hospital.
Who Masked: Outcomes Assessor
Masking Description: It will not be possible to mask for either patients nor participating health care professionals if patients are enrolled in the control- or intervention group. Hence, the study will not be blinded. When the final data analysis is performed for the primary outcome measure the person performing the analysis will not be aware of which group each patient was a part of.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MRI group (Experimental): An abbreviated MRI of the liver/abdomen
  Interventions: Radiation: Abbreviated MRI of the liver/abdomen
- CT group (Active Comparator): A combined single venous and 3 min equilibrium phase CT of the abdomen/liver
  Interventions: Radiation: Combined single venous and 3 min equilibrium phase CT of the abdomen/liver

INTERVENTIONS:
Radiation: Abbreviated MRI of the liver/abdomen — The MRI examinations of the liver/abdomen will be performed at the same time as the pelvic MRI. A 1,5 T scanner will be used together with a dedicated torso/abdominal coil. An abbreviated MRI liver protocol includes 3 different sequences as follows:
  1. Axial T2-weighted respiratory triggered sequence with 5 mm slice thickness.
  2. Axial diffusion weighted spin echo respiratory triggered sequence with fatsat with b-factors 50/800 s/mm2 and ADC calculation maps, 5 mm slice thickness
  3. An axial breath-hold 3D T1-weighted gradient echo with fatsat with 4 mm slice thickness, gap 2 mm, contrast enhanced venous phase and in a 3 min equilibrium phase, using regular i.v bolus injection of gadolinium contrast medium with standard clinical dose.
  Arms: MRI group
Radiation: Combined single venous and 3 min equilibrium phase CT of the abdomen/liver — The CT examination of the liver will be performed as a combined examination in a single venous phase starting with the thoracic region directly followed by the abdomen down to the pelvis. An additional 3 min equilibrium phase of the liver only will end the examination. Regular iodinated low-osmolar non-ionic contrast media will be used of 350 mg I/ml using a power injector, 2-4 ml/s, 100-150 ml dependent on patient weight and kidney function. Reconstructed images in axial, coronal and sagittal plane will be performed.
  Arms: CT group

SUMMARY:
This multicentre randomized controlled trial aims to investigate whether an abbreviated MRI is comparable to a combined single venous phase CT with an additional 3 min equilibrium phase of the liver, in the pretreatment radiological workup in patients with rectal cancer.

DETAILED DESCRIPTION:
The incidence of rectal cancer in the European Union is approximately 125 000 per year, constituting a third of the total colorectal cancer incidence(1). In Sweden approximately 2000 individuals are diagnosed with rectal cancer each year. Evaluation of patients and possible treatment strategies (including neo-adjuvant chemo/radiotherapy, choice of surgical technique and adjuvant chemotherapy) are based on tumor specific characteristics together with patient factors such as general condition and comorbidity. These characteristics include tumor, lymph node and metastasis classification (cTNM), height of tumor (distance from anal verge), engagement of circumferential margin or mesorectal fascia, signs of extramural invasion and the presence of distant metastases. Clinical examination and endoscopy together with magnetic resonance imaging (MRI) of the pelvic region are essential in the local staging process, where MRI provides the most accurate radiological assessment, especially for rectal tumors in stage T3 and T4. The recommended methods regarding evaluation of metastases (M stage) include contrast enhanced computed tomography (CT) or MRI of the liver/abdomen, CT of the thorax, and in selected cases positron emission tomography (PET)- CT, if extensive extramural vascular invasion is present.

Previous studies have investigated the efficiency of MRI compared to other radiological methods and found that MRI of the liver is superior to contrast enhanced CT, in terms of specificity and sensitivity for diagnosis of liver metastasis (both per patient and per lesion).

Even though MRI has been recommended as the first line modality for evaluating colorectal cancer liver metastases in patients who have not previously undergone therapy the Swedish national guidelines, as well as the European Society for Medical Oncology (ESMO), include recommendations of single venous phased contrast enhanced CT of the liver/abdomen in the pre-treatment radiological workup. Progress within diagnostics has led to development of CT examination with an additional 3 min equilibrium phase of the liver that may be added to the single venous phase in order to increase the sensitivity and specificity of the diagnosis of liver metastases. However, this has not yet been included in guidelines nor implemented on a national basis in the pre-treatment radiological workup in patients with colorectal cancer.

Objective The primary objective of the present study is to compare percentage of patients requiring further radiological examinations after index examination (due to inconclusive results) between patients randomized to an abbreviated MRI liver protocol and patients randomized to a combined single venous phase CT with an additional 3 min equilibrium phase of the liver. A secondary aim is to compare time to treatment initiation, survival and development of liver metatstases between patients randomized to either an abbreviated MRI or a combined single-venous phase CT with an additional 3 min equilibrium phase of the liver.

The study is a multicentre randomized controlled trial where the hypothesis is that there is no clinical difference between the two groups, and the study is designed as a non inferiority trial.

ELIGIBILITY:
Inclusion Criteria:

* Adults >18 years of age
* Endoscopically or clinically diagnosed with (suspected) rectal cancer and considered for further radiological investigation
* Are able to understand trial information and provide oral and written consent

Exclusion Criteria:

* Patients unable to undergo MRI (causes may include claustrophobia, presence of pacemaker or certain metal components in their body).
* Patients diagnosed with benign disease of the rectum or squamous cell carcinoma
* Patients diagnosed with recurrent rectal cancer
* Patients unable to understand the trial information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2022-04-12 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Need for supplementary radiologic liver examination | 3 months
  Number of patients in need for supplementary radiologic liver examination/s before treatment decision, after index examination (CT or MRI) of the abdominal organs, due to inconclusive results.
Cost effectiveness | 12 months
  Costs related to all index radiological examinations will be included. Costs will be collected from national sources such as the Swedish association of local authorities and regions (SKR - Sveriges kommuner och regioner) whenever possible and alternatively from Sahlgrenska university hospital cost-per-patient files. Possibly a more complex model will be relevant depending on outcome, where total health care costs are compared between the two radiological work-up routines. Such an analysis will take survival into account.

SECONDARY OUTCOMES:
Time to start of treatment | 12 months
  Time from index radiological workup to start of treatment
Recurrence of rectal cancer | 12 months
  Number of patients with recurrence of rectal cancer (local or metastatic disease)
Liver metastasis | 36 months
  Number of patients diagnosed with liver metastasis
Survival | 36 months
  Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Park, MD, PhD, Principal Investigator — Sahlgrenska University Hospital, Sahlgrenska Academy, Gothenburg Sweden
Locations (1):
- Sahlgrenska University Hospital/Östra, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Van Cutsem E, Cervantes A, Adam R, Sobrero A, Van Krieken JH, Aderka D, Aranda Aguilar E, Bardelli A, Benson A, Bodoky G, Ciardiello F, D'Hoore A, Diaz-Rubio E, Douillard JY, Ducreux M, Falcone A, Grothey A, Gruenberger T, Haustermans K, Heinemann V, Hoff P, Kohne CH, Labianca R, Laurent-Puig P, Ma B, Maughan T, Muro K, Normanno N, Osterlund P, Oyen WJ, Papamichael D, Pentheroudakis G, Pfeiffer P, Price TJ, Punt C, Ricke J, Roth A, Salazar R, Scheithauer W, Schmoll HJ, Tabernero J, Taieb J, Tejpar S, Wasan H, Yoshino T, Zaanan A, Arnold D. ESMO consensus guidelines for the management of patients with metastatic colorectal cancer. Ann Oncol. 2016 Aug;27(8):1386-422. doi: 10.1093/annonc/mdw235. Epub 2016 Jul 5. PMID 27380959
- [Background] Achiam MP, Logager VB, Skjoldbye B, Moller JM, Lorenzen T, Rasmussen VL, Thomsen HS, Mollerup TH, Okholm C, Rosenberg J. Preoperative CT versus diffusion weighted magnetic resonance imaging of the liver in patients with rectal cancer; a prospective randomized trial. PeerJ. 2016 Jan 14;4:e1532. doi: 10.7717/peerj.1532. eCollection 2016. PMID 26793420
- [Background] Niekel MC, Bipat S, Stoker J. Diagnostic imaging of colorectal liver metastases with CT, MR imaging, FDG PET, and/or FDG PET/CT: a meta-analysis of prospective studies including patients who have not previously undergone treatment. Radiology. 2010 Dec;257(3):674-84. doi: 10.1148/radiol.10100729. Epub 2010 Sep 9. PMID 20829538
- [Background] Ferlay J, Steliarova-Foucher E, Lortet-Tieulent J, Rosso S, Coebergh JW, Comber H, Forman D, Bray F. Cancer incidence and mortality patterns in Europe: estimates for 40 countries in 2012. Eur J Cancer. 2013 Apr;49(6):1374-403. doi: 10.1016/j.ejca.2012.12.027. Epub 2013 Feb 26. PMID 23485231
- See also: National Cancer Care Guidelines for Colorectal Cancer [National Cancer Care Guidelines]. — http://www.cancercentrum.se